CLINICAL TRIAL: NCT05205148
Title: Ultrathin Drug Eluting Stents for Patients With Left-main, bifurcaTion, chRonic totAl Occlusion, or In-stent Restenosis Coronary Lesion in Real Life: the ULTRA a Multicenter Study
Brief Title: Ultrathin DES in Complex PCI Scenarios: the ULTRA a Multicenter Study
Acronym: ULTRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Fabrizio D'Ascenzo, Clinical Professor, A.O.U. Città della Salute e della Scienza
Other Study IDs: ULTRA registry
Record Dates: First submitted 2022-01-05; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Disease; Coronary Stenosis; Stent Restenosis; Left Main Coronary Artery Disease; Chronic Total Occlusion of Coronary Artery
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Percutaneous coronary intervention with the following platforms: Orsiro; Mistent; BioMime; Supraflex Cruz — Patients treated with ultrathin coronary stents (namely stents with strut thickness < 70 um) for specific coronary disease scenarios: unprotected left main stenosis; Bifurcation coronary stenosis (with side branch diameter ≥ 2.5 mm); Chronic total coronary occlusion; In-stent restenosis

SUMMARY:
ULTRA is a multicenter, observational, retrospective registry, enrolling consecutive patients treated with ultrathin coronary DES (coronary stent with strut thickness < 70 um) for coronary bifurcation lesions, left main disease, chronic total coronary occlusion, and in-stent restenosis regardless of their clinical presentation. Target lesion failure (TLF a composite endpoint of cardiovascular death, target vessel myocardial infarction, target lesion revascularization and definite stent thrombosis) will be the primary end point, while its single components will be the secondary ones along with all-cause death, all acute myocardial infarction (excluding peri-procedural AMI), target vessel revascularization and BARC major bleedings (BARC 3-5). Due to the retrospective, observational nature of the registry, no formal sample size estimation is required. Patients complying with detailed inclusion criteria and with a minimum follow up of 6 months will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* Unprotected left main stenosis
* Bifurcation coronary stenosis (with side branch diameter ≥ 2.5 mm)
* Chronic total coronary occlusion
* In-stent restenosis

Treated with the following devices:

* Orsiro
* Mistent
* BioMime
* Supraflex Cruz

Exclusion Criteria:

* patients died during the index revascularization procedure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients treated with ultrathin coronary DES for coronary bifurcation lesions, left main disease, chronic total coronary occlusion and in-stent restenosis regardless of their clinical presentation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of target lesion failure (TLF) | Up to 2 years
  A composite endpoint of cardiovascular death, target vessel myocardial infarction, target lesion revascularization and definite stent thrombosis

SECONDARY OUTCOMES:
Incidence of all-cause death | Up to 2 years
  death from any cause
Incidence of acute myocardial infarction (AMI) | Up to 2 years
  all acute myocardial infarction excluding peri-procedural myocardial infarction
Incidence of target vessel revascularization (TVR) | Up to 2 years
  All revascularization in a vessel treated with ultrathin DES within the index procedure
Incidence of major bleedings | Up to 2 years
  Major bleedings defined according to Bleeding Academic Research Consortium (BARC 3-5)
Incidence of cardiovascular death | Up to 2 years
  Death from cardiovascular causes
Incidence of target Vessel Myocardial Infarction | Up to 2 years
  Myocardial infarction whose culprit artery is unequivocally identified as an artery treated with ultrathin Drug eluting stent within the index procedure
Incidence of target lesion revascularization | Up to 2 years
  coronary revascularization due to acute coronary syndrome or stable ischemic presentation due to a lesion previously treated with ultrathin drug eluting stent within the index procedure
Incidence of definite stent thrombosis | Up to 2 years
  stent thrombosis in a coronary segment previously treated with ultrathin drug eluting stent

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio D'Ascenzo, PhD, Principal Investigator — AOU Città della Salute e della Scienza Torino
Locations (1):
- Fabrizio D'Ascenzo, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi KH, Nam CW, Bruno F, Cho YK, De Luca L, Kang J, Mattesini A, Song YB, Truffa A, Kim HS, Wanha W, Chun WJ, Gili S, Helft G, Han SH, Cortese B, Lee CH, Escaned J, Yoon HJ, Chieffo A, Hahn JY, Gallone G, Choi SH, De Ferrari G, Koo BK, Quadri G, Hur SH, D'Ascenzo F, Gwon HC, de Filippo O. Differential Prognosis of True Bifurcation Lesions According to Left Main Versus Non-Left Main Location and Treatment Strategy. J Am Heart Assoc. 2025 Feb 4;14(3):e037657. doi: 10.1161/JAHA.124.037657. Epub 2025 Feb 3. PMID 39895551
- [Derived] De Filippo O, Wanha W, Sanavia T, Januszek R, Giacobbe F, Campo G, Pinxterhuis TH, Capodanno D, Tomasiewicz B, Iannaccone M, Leone A, Wolny R, Bruno F, Patti G, Musumeci G, Liccardo G, Verardi R, Roubin SR, Tarantini G, Kuzma L, Perl L, Gagnor A, Reczuch K, Conrotto F, Tuttolomondo D, Ploumen EH, Niezgoda P, Caglioni S, Omede P, Greco A, Kubica J, Gil RJ, Piccolo R, Kornowski R, Bil J, Morena A, Zocca P, Pennone M, Gasior M, Jaguszewski M, von Birgelen C, Fariselli P, De Ferrari GM, Wojakowski W, D'Ascenzo F. Treatment of in-stent restenosis with ultrathin-strut versus thin-strut drug-eluting stents or drug-eluting balloons: a multicentre registry. EuroIntervention. 2024 Nov 4;20(21):e1340-e1354. doi: 10.4244/EIJ-D-24-00491. PMID 39492702